CLINICAL TRIAL: NCT04431622
Title: Objective Measurement of Hearing Aid Benefit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study did not receive funding
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Samira Anderson, Associate Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 415685-15
Record Dates: First submitted 2020-03-17; First posted 2020-06-16 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Auditory Perceptual Disorders; Age-related Hearing Loss
MeSH Terms: conditions — Auditory Perceptual Disorders; Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effects of hearing aid algorithms (Experimental): Neural processing and cognitive effort will be assessed in individuals who listen to stimuli generated with linear and fast-acting compression hearing aid algorithms and with actual hearing aids.
  Interventions: Device: Hearing aid amplification algorithms

INTERVENTIONS:
Device: Hearing aid amplification algorithms — The investigators will use stimulus waveforms that have been amplified and recorded for each individual's hearing loss. These waveforms will be created using Desired Sensation Level, Version 5-C hearing aid targets on a continuum of increased signal manipulation. The NIH-funded open hearing aid platform will be used to provide precise control over hearing aid parameters to create waveforms with linear and fast-acting compression amplification. A third set of waveforms will be created using a current clinical hearing aid that uses typical noise reduction and compression parameters. Investigating the effects of hearing aid algorithms in young normal-hearing and older normal-hearing listeners will aid in interpretation of these effects in the older hearing-impaired listeners.

SUMMARY:
Hearing loss is a critical health concern in the rapidly aging population, affecting approximately 22 million older individuals in the United States. Yet, only 30% of individuals who would benefit from the use of hearing aids regularly use them. This project aims to improve the benefit of hearing aids for older adults through incorporation of objective neural measures to assess effects of hearing aid algorithms.

DETAILED DESCRIPTION:
Hearing loss is among the top three major health conditions in older adults and has been identified as a major modifiable risk factor for dementia. It is therefore imperative that older adults receive effective treatment for hearing loss in a timely manner to prevent losses in social, emotional, and cognitive function. The current hearing aid fitting is based on audiometric thresholds, but this approach does not account for large individual differences in auditory temporal perception and cognitive ability that may affect speech understanding in challenging listening environments. At present, there is a gap in knowledge of how best to fit hearing aids for individual listeners. The long-term goal is to improve the benefit of hearing aids for older adults so that they can maintain independence and quality of life. The overall objective of this proposal is to identify the neural temporal processing mechanisms associated with individual differences in hearing aid benefit in older adults with similar audiograms. The investigators will use the innovative approach of combining complementary neural and behavioral measures to assess the effects of hearing aid amplification on speech perception and effortful listening. The central hypothesis is that the neural representation of the temporal envelope of speech can be used to predict hearing aid benefit in older adults with hearing loss. The central hypothesis will be tested through the pursuit of three aims: (1) Measure the extent to which amplification distorts the neural and perceptual processing of temporal cues; (2) Quantify reductions in temporal envelope tracking and increases in cognitive effort associated with amplification algorithms that distort the temporal envelope of the speech signal; and (3) Investigate the use of objective physiological measures of temporal processing to predict hearing aid benefit. The expected outcome is the development of an objective, neurophysiological tool for use in the design and fitting of advanced algorithms to maximize speech perception in a variety of listening environments. This outcome is expected to have a positive impact on the treatment of hearing loss and its sequelae in older adults, because it will lead to a better understanding of the neural mechanisms contributing to successful use of hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Aims 1 and 2 age ranges: 18-35 and 60-75
* Aim 3 age range: 50 to 85
* Aims 1 and 2 hearing levels: 1) Normal hearing thresholds defined as pure-tone thresholds ≤ 20 decibel (dB) hearing level (HL) from 125 to 4000 Hz and ≤ 30 dB HL at 6000 and 8000 Hz bilaterally, or 2) Mild to moderate sensorineural hearing loss defined as thresholds within 5 dB of 30 dB HL at 500 Hz, 50 dB HL at 1000 and 2000 Hz, and 60 dB HL at 4000 Hz.
* Aim 3 hearing level: Symmetric hearing thresholds with no interaural difference ≥ 15 dB HL at ≥ 2 frequencies.
* Intelligent Quotients ≥ 85 based on the Wechsler Abbreviated Scale of Intelligence (Psychological Corp., New York)
* Scores ≥ 24 on the Montreal Cognitive Assessment

Exclusion Criteria:

* Neurological disorders
* Middle ear pathology
* Nonnative English speakers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Neural response fidelity | Immediately post-treatment
  Neuroelectric and neuromagnetic responses are recorded to amplified one-minute speech samples. Reconstruction of the speech envelope will be performed using a linear reconstruction matrix estimated via boosting. Reconstruction success is measured by the linear correlation between the reconstructed and the acoustic speech envelope.

SECONDARY OUTCOMES:
Cognitive effort | Immediately post-treatment
  Cognitive effort is inferred from pupillometry data Growth-curve analysis will be used to determine pupil response amplitude.

IPD SHARING:
Plan to Share IPD: Yes
Publication of data and other research products shall occur during the project, if appropriate, or at the end of the project, consistent with practices in our field. De-identified data that document, support, and validate research findings will be made available when the main findings have been accepted for publication. Research products from this project will be archived at the Digital Repository at the University of Maryland (DRUM) unless a more appropriate facility can be identified. DRUM is a long-term, open access repository managed and maintained by the University of Maryland Libraries. Researchers and the general public can download data and code files, associated metadata and documentation, and any guidelines for reuse. All records in DRUM are assigned a persistent Digital Object Identifier (DOI) to support consistent discovery and citation. The project description will be automatically indexed in Google Scholar to support global discovery.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available at the end of the project for an indefinite period.
Access Criteria: For the research products available to the public, there are no conditions on reuse or redistribution beyond the attribution and credit norms of the scientific community. In the event that reviewers or researchers wish to examine data containing direct or indirect identifiers, they will be required to conform to the terms of a data use agreement. The agreement will prohibit redistribution of sensitive data.